CLINICAL TRIAL: NCT04821427
Title: Feasibility of an mHealth + Brief Intervention for Heavy Drinking African American and Latino MSM: A Pilot Study
Brief Title: Alcohol and Sex Risk mHealth-Enhanced Brief Intervention for BLMSM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Kathryn Chavez, Clinical Psychology Doctoral Candidate, Department of Psychological and Brain Sciences, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5479E
Record Dates: First submitted 2021-03-23; First posted 2021-03-29 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Heavy Drinking and Sexual Risk Behavior
Keywords: heavy drinking; sexual risk behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief mHealth Intervention + mobile messaging (Experimental): The intervention is a brief, motivational video-conferencing intervention followed by four weeks of app-based, interactive mobile messages
  Interventions: Behavioral: Brief mhealth intervention + mobile messaging to reduce sexual risk behavior and heavy drinking
- Assessment Only (No Intervention): This is an assessment only condition. No intervention following completion of baseline surveys will be administered.

INTERVENTIONS:
Behavioral: Brief mhealth intervention + mobile messaging to reduce sexual risk behavior and heavy drinking — The intervention is a brief, motivational video-conferencing intervention followed by four weeks of app-based, interactive mobile messages to reduce heavy episodic drinking and sexual risk behavior (condomless anal intercourse) among Black/African American and Hispanic/Latino men who have sex with men
  Arms: Brief mHealth Intervention + mobile messaging

SUMMARY:
Randomized controlled pilot trial to test the feasibility and efficacy of a brief intervention with app-based messaging to reduce sexual risk behavior and heavy drinking among Black/African American and Hispanic/Latino MSM.

DETAILED DESCRIPTION:
This study seeks to develop and provide an initial test of a brief intervention to reduce alcohol use and sex risk behavior among Black and Latino men who have sex with men [BLMSM]. The study seeks to recruit BLMSM who are non-monogamous, not currently on pre-exposure prophylaxis [PrEP], have engaged in condomless anal intercourse over the past 6 months, who have engaged in heavy drinking defined as >14 drinks per week or at least 1 heavy drinking episode (5+ drinks on a single occasion) in the past month. All participants will complete baseline measures about past month behavior and if eligible will be assigned to the intervention condition or an assessment only condition. The intervention consists of a single brief video-conferencing intervention coupled with 4 weeks of mobile-messaging related to individualized goals about alcohol use and sexual behavior. Follow-up assessments are scheduled for 4 weeks after baseline (upon completion of the mobile-messaging component of the intervention) and 2 months after baseline. Primary outcomes are feasibility and acceptability of the intervention and mobile-messaging components. Secondary outcomes are changes in frequency of condomless anal intercourse and heavy drinking episodes.

ELIGIBILITY:
Inclusion Criteria:

* Black/African American or Latino/Hispanic
* At least one heavy drinking episode in past month
* At least one episode of condomless anal intercourse with another man in the past 6 months
* Own a smartphone
* English speaking

Exclusion Criteria:

* HIV+
* Currently on PrEP
* Monogamous/exclusive relationship
* Past or current treatment for alcohol (past 3 years)
* Current or past psychiatric treatment (past 3 months)
* Diagnosis of Bipolar Disorder or Schizophrenia
* Brief Michigan Alcoholism Screening Test score >5
* Lifetime diagnosis of substance use disorder
* ASSIST score of >/=27 for any individual substance

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Modified Daily Drinking Questionnaire - Heavy Drinking Episodes | Past 30 days
  Number of heavy drinking episodes NIAAA criteria (5+ drinks)
Sexual Behavior - Extended Survey - Condomless Anal Intercourse | Past 30 days
  Frequency of condomless anal intercourse. This is an open ended question where the Participant reports the frequency of condomless anal intercourse over the past 30 days.

SECONDARY OUTCOMES:
Goal Systems Assessment Battery - Alcohol | Past 30 days
  Ratings of self-regulatory capacities related to reducing alcohol use. Items are 5-point Likert scale. There are 4 subscales utilized including planning, monitoring, self-efficacy and value. Higher scores indicates better outcomes.
Goal Systems Assessment Battery - Condom Use | Past 30 days
  Ratings of self-regulatory capacities related to using condoms. Items are 5-point Likert scale. There are 4 subscales utilized including planning, monitoring, self-efficacy and value. Higher scores indicates better outcomes.
Client Satisfaction Questionnaire | 2 months post-baseline
  8-item Client Satisfaction Questionnaire answered on a 4-point scale. Mean scale score is 1-4. Higher scores reflect a better outcome.
Intervention Acceptability Ratings | 2 months post-baseline
  10-item Acceptability Measure of the overall intervention answered on a 5-point Likert scale (strongly disagree to strongly agree) used to assess the acceptability of the video-conferencing brief intervention and the mobile messages. Mean scale range is 1-5. Higher scores reflect a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn E Chavez, MA, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
under discussion